CLINICAL TRIAL: NCT00924976
Title: Improving Representative Payeeship for People With Psychiatric Disabilities and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: H133G070058
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2011-05

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects will be offered the Steps for Achieving Financial Empowerment (SAFE) which helps facilitate a cooperative consumer-payee relationship, increase accurate knowledge about representative payeeship, promote collaborative money management and effective budgeting, and prepare mutually developed plans for carrying out the payeeship in the future.
  Interventions: Behavioral: Steps for Achieving Financial Empowerment (SAFE)
- 2 (No Intervention): Representative payeeship as usual

INTERVENTIONS:
Behavioral: Steps for Achieving Financial Empowerment (SAFE) — The SAFE is a brief, 5-component intervention that aims to facilitate a cooperative consumer-payee relationship, increase accurate knowledge about representative payeeship, promote collaborative money management and effective budgeting, and prepare mutually developed plans for carrying out the payeeship in the future.
  Arms: 1

SUMMARY:
Representative payees, mostly family members, manage Social Security Administration funds of more than one million people with psychiatric disabilities. Although studies show payeeship can be used coercively, foster dependency, reduce work incentives, lead to family conflict and even violence, there has been little systematic research on how to lower these significant barriers to community integration.

The investigators' long term goal is to promote recovery among adults with psychiatric disabilities who have payees by reducing downsides associated with what has been called "the nation's largest guardianship system." The investigators' objective in the current application is to evaluate a pilot-tested, stakeholder-informed intervention that is grounded in principles of psychiatric rehabilitation and encourages consumers with psychiatric disabilities and their family members to collaborate within the representative payee arrangement.

DETAILED DESCRIPTION:
To do this, we will test the Steps for Achieving Financial Empowerment (SAFE) intervention by randomly assigning N=200 consumer-family payee dyads into one of two groups: (a) the SAFE intervention (n=100); or (b) a "usual care" control (n=100). The SAFE is a brief, 5 component educational intervention that aims to facilitate a cooperative consumer-payee relationship, increase accurate knowledge about representative payeeship, promote collaborative money management and effective budgeting, and prepare mutually developed plans for carrying out the payeeship in the future.

We will interview people with psychiatric disabilities and their family payees at baseline and six-months. This study aims to examine the effects of the SAFE intervention on community participation, employment, and family support of adults with psychiatric disabilities who have family representative payees. Our central hypothesis, based on strong preliminary data, is that the SAFE will benefit consumers by enhancing autonomy, boosting motivation to work, and reducing family conflict.

ELIGIBILITY:
Inclusion Criteria:

* For disability recipients:

  1. Meets DSM-IV criteria for schizophrenia, schizoaffective disorder, bipolar disorder, or depressive disorder with psychotic features;
  2. age 18-65;
  3. Has a family member (parent or sibling) as a representative payee.
* For payees:

  1. Has family member (child or sibling) with schizophrenia, schizoaffective disorder, bipolar disorder, or depressive disorder with psychotic features; and
  2. Is the family member's representative payee.

Exclusion Criteria:

* None.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2008-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
employment | six months
empowerment | six months
family support | six months

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Elbogen, Ph.D., Principal Investigator — UNC-Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Elbogen EB, Ferron JC, Swartz MS, Wilder CM, Swanson JW, Wagner HR. Characteristics of representative payeeship involving families of beneficiaries with psychiatric disabilities. Psychiatr Serv. 2007 Nov;58(11):1433-40. doi: 10.1176/ps.2007.58.11.1433. PMID 17978253
- [Background] Elbogen EB, Wilder C, Swartz MS, Swanson JW. Caregivers as money managers for adults with severe mental illness: how treatment providers can help. Acad Psychiatry. 2008 Mar-Apr;32(2):104-10. doi: 10.1176/appi.ap.32.2.104. PMID 18349329
- [Background] Elbogen EB, Tiegreen J, Vaughan C, Bradford DW. Money management, mental health, and psychiatric disability: a recovery-oriented model for improving financial skills. Psychiatr Rehabil J. 2011 Winter;34(3):223-31. doi: 10.2975/34.3.2011.223.231. PMID 21208861